CLINICAL TRIAL: NCT05464992
Title: Use of CEST (Chemical Exchange Saturation Transfer) Imaging in PET/MRI
Acronym: GlioCEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-005; 2022-A00910-43 (Other: ID-RCB Number)
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Glioma; Brain Metastases
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with glioma or brain metastases (Other)
  Interventions: Other: Additional CEST sequences during PET/MRI exam

INTERVENTIONS:
Other: Additional CEST sequences during PET/MRI exam — CE-Marked Advanced Technology Software Modules (ATSM) for Magnetic Resonance Imaging from General Electric Healthcare

SUMMARY:
Standard Magnetic Resonance Imaging (MRI) is based on the excitation of hydrogen nuclei that are presents in water molecules, which abundance in human body allows for obtention of superior contrast. However, assessing the presence of other molecules than water in tissues is also of great clinical interest to probe metabolites related to physiological body function and pathological conditions.

Chemical exchange saturation transfer (CEST) allow to overcome some limitations of proton magnetic resonance spectroscopy (1H-MRS) by exploiting chemical properties of the targeted molecule through a continuous process of re-saturation and exchange, and thus detecting it with increased sensitivity, from two orders of magnitude. Moreover, CEST technique is based on imaging sequences and can therefore benefit from well-known fast acquisition strategies, as well as improved spatial resolution.

DETAILED DESCRIPTION:
For this study the investigators propose to include an additional CEST sequence in standard PET/MRI exam in order to obtain a cartography with biochemical informations from tissues in patients with glioma or brain metastases.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the Nuclear Medicine and Molecular Imaging department of ICANS (Institut de cancérologie strasbourg Europe) for a PET/MRI exam dedicated to:

* Preoperative evaluation of a cerebral expansion lesion
* Evaluation of glioma recurrences
* Evaluation of brain metastases
* Evaluation of recurrence of metastases

Exclusion Criteria:

* Contraindication to the realization of an MRI
* Minor or patients placed under guardianship or supervision
* Patients deprived of liberty
* Patients placed under judicial protection
* Patients that are not able to express their consent
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2036-12-28 (Estimated); Study Completion 2036-12-28 (Estimated)

PRIMARY OUTCOMES:
Obtention, from a set of brain PET-MRI images, of an intratissular pH mapping in patients with glioma or brain metastases | through study completion, up to 14 years
  Evaluation at the cerebral level on the acquisition images of residual volume in MRI
Obtention, from a set of brain PET-MRI images, of an intratissular pH mapping in patients with glioma or brain metastases | through study completion, up to 14 years
  Evaluation at the cerebral level on the acquisition images of tumoral metabolic activity in PET

SECONDARY OUTCOMES:
Correlate intratissular pH mapping and location of recurrence | through study follow-up, up to 10 years
Correlate average pH of the tumor and histopathology | through study follow-up, up to 10 years
Correlate average pH of the tumor and Disease-Free Survival (DFS) | through study follow-up, up to 10 years
Correlate average pH of the tumor and Overall survival (OS) | through study follow-up, up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- France Institut de cancérologie Strasbourg Europe, Strasbourg, France